CLINICAL TRIAL: NCT05219890
Title: Longitudinal Analysis of the Transcriptome From Mononuclear Blood Cells and of the Inflammatory Status of Obese Patients, Supplemented With High Doses of Omega-3 Fatty Acids (EPA and DHA)
Brief Title: Transcriptomics of Mononuclear Cells and Inflammatory Status of Obese Patients Treated With Omega-3 Fatty Acids
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We reached the number of participants required.
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1832
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-01

CONDITIONS: Obesity; Inflammation; Immune System Disorder
Keywords: omega-3 fatty acids; DHA; EPA
MeSH Terms: conditions — Obesity; Inflammation; Immune System Diseases | interventions — Fish Oils

STUDY DESIGN:
Intervention Model Description: Healthy volunteers and obese patients will consume the same amount of omega-3 fatty acids for the same time.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OBESE PATIENTS (Experimental): Obese patients will be recruited from the outpatient Clinic of Obesity at the INCMNSZ. They will consume the fish oil equivalent to 4.8 g/day of EPA and DHA for 3 months, followed by a one-month period without treatment.
  Interventions: Dietary Supplement: Fish oil
- CONTROL GROUP (Active Comparator): Healthy normal volunteers will be recruited from friends and family of the investigators, and staff at the INCMNSZ. They will consume the fish oil equivalent to 4.8 g/day of EPA and DHA for 3 months, followed by a one-month period without treatment.
  Interventions: Dietary Supplement: Fish oil

INTERVENTIONS:
Dietary Supplement: Fish oil — They will consume the fish oil equivalent to 4.8 g/day of EPA and DHA for 3 months, followed by a one-month period without treatment.

SUMMARY:
The main objective is to determine the effect that supplementation with 4.8 g/day of w-3 FA [3.2g eicosapentaenoic acid (EPA) and 1.6 g docosahexaenoic acid (DHA)] have on the inflammatory state of obese patients (BMI ≥ 35.0 kg/m2), at the metabolic, cellular and molecular levels.

DETAILED DESCRIPTION:
Methodology Study design. This is a prospective, experimental, comparative, non-blinded (open) study.

Adult obese (BMI ≥ 35.0 kg/m2) patients, age 25 to 45 y, of any gender will be recruited from the outpatient Clinic of Obesity at the INCMNSZ. The patients may have (or not) insulin resistance, but must not have any of the following: type 2 diabetes (controlled or not), hypertension, liver or kidney failure, metabolic syndrome, taking antinflammatory drugs or dietary supplements, and in the case of women, pregnant or lactating.

The control group will consist of 40 healthy adult non-obese volunteers (BMI 18.5 to 23.0 kg/m2), age 25 to 45 y, of any gender who accept to participate in the study. This group will only be studied at the beginning (time 0) and they will not consume the fish oil supplement, since its use will be to obtain reference values for all variables described.

Fish oil supplement will be the source of omega-3 fatty acids (w-3 FA) and this will be a donation from the Inflammation Research Foundation (IRF, Boston MA), in the form of sealed unmarked bottles with 120 capsules/bottle.

Each 1 gram capsule contains 0.6 g of w-3 FA (0.4 g of EPA and 0.2 g of DHA). In order to provide 4.8 g of w-3 FA each obese patient must consume 8 capsules/day, distributed as follows: 2 capsules at breakfast, 4 capsules with the main meal and 2 capsules at dinner.

Study design. Each participant (control subjects and obese patients) will receive 2 bottles (240 capsules) of the fish oil at the time of recruitment (time 0) which is enough to cover the dosage for 1 month. After the first month had passed, the remaining capsules (if any) will be counted and 2 new bottles of supplement will be provided to cover the dosage of the following month. This strategy will be repeated at the end of month +2 to cover the dosage of month +3. A "wash-out" period of at least 1 month will be observed (month +4). All variables described (except anthropometry) will be analyzed at times 0, +2 and +4.

Anthropometry. Height in meters (m), weight in kilograms (kg), will be used to calculate the body mass index (BMI) with the formula [weight (kg)/ height (m)2]. Body composition will be determined by electric bioimpedance with a Full Body Composition Analyzer X-Contact 356, to quantify the fat mass (in % and in kg) and the fat-free (lean) mass (in % and kg). Anthropometry will be done only at times 0 and +4.

Blood samples. Venous blood will be obtained at times 0, +1, +2, +3 and +4 with the Vacutainer system with anticoagulant (EDTA-K2). An aliquot of blood will be centrifuged to obtain plasma and stored at -80°C until assayed. Peripheral blood mononuclear cells (PBMNC) will be obtained by density gradient centrifugation (Lymphoprep). These cells will be further processed for the following determinations: i) transcriptional analysis by RNA-seq and qPCR, ii) flow cytometry analysis of immune cells populations (B, T and monocytes), iii) cellular and energy metabolism (Seahorse) and, iv) the "Treg-mediated suppression of cellular proliferation (TMSCP)" assay.

Biochemical analysis. Serum levels of the following metabolites, lipids, cytokines and adipokines will be determined: glucose, insulin, total cholesterol, HDL, LDL, triglycerides, adipokines (leptin, adiponectin, IL-6, TNFalpha, MCP1), and interleukin (IL) 1beta, 2, 4, 8, 10, 12, 17 and TGFbeta. Fatty acid levels will be determined by gas chromatography in serum samples, and in cellular membranes from erythrocytes and leukocytes (PBMNC). The concentration of SPM (resolvins, protectins and maresins) will be determined by HPLC coupled to a mass spectrometer.

Bioenergetics analysis of PBMNC. Cellular metabolism will be analyzed with a Seahorse XFe96 Analyzer (Agilent) to measure oxygen consumption rate (OCR) and extracellular acidification rate (ECAR) of live cells in a 96-well plate format. OCR and ECAR rates are key indicators of mitochondrial respiration and glycolysis respectively. From this analysis of energy consumption, a "bioenergetic health index" (BHI) will be obtained. This BHI reflects the dominant source of energy employed by the cells and can reflect the metabolic pathway employed. For instance, if a high amount of OCR is obtained, this reflects an aerobic metabolism (fatty acid oxidation and oxidative phosporylation, ie, FAO and OXPHOS), whereas a high ECAR indicates anaerobic metabolism and glycolysis is the main metabolic pathway employed.

Transcriptional analysis of gene expression. Total RNA will be obtained from PBMNC and subpopulations (namely, monocytes and Treg cells) using the Trizol reagent and isopropanol precipitation. RNA integrity will be determined in 1% agarose gels by electrophoresis and its concentration by UV spectrophotometry at 260nm.

Samples of RNA with RIN values of 8 and higher will used for sequencing; complementary DNA (cDNA) will be synthesized with reverse-transcriptase and (dT)15 oligonucleotides. The ends of the cDNA fragments will be ligated to sequencing adaptors and amplified by PCR to produce the RNA-Seq library, which will be ready for sequencing. The sequencing method used in the present study will be next generation sequencing (NGS) with the Illumina platform. Validation of changes in the level of transcription determined by RNA-seq analysis, will be determined by quantitative real-time polymerase chain reaction (qPCR) using a RotorGeneQ thermocycler and SybrGreen as label. 18S rRNA will be used as housekeeping gene.

The most powerful use of RNA-Seq is finding differences in gene expression between two or more conditions (e.g., obese vs not obese); this process is called differential expression. The outputs are frequently referred to as differentially expressed genes (DEGs) and these genes can either be up- or down-regulated (i.e., higher or lower in the condition of interest). A cut-off point of 2 fold difference with a p value <0.05 may be used as a screening procedure (although more astringent thresholds may be applied) followed by graphic resources (volcano plots and a heat maps) that will allow identification of transcripts with the largest expression differences and significance. The list of differentially expressed genes will be analyzed using KEGG, IPA and/or Metacore to predict which metabolic/biochemical process differ between the obese and control groups, and after the supplement with fish oil in the obese group.

ELIGIBILITY:
Inclusion Criteria:

Control group:

* healthy adult non-obese volunteers (BMI 18.5 to 23.0 kg/m2)

Obese group:

* metabolically healthy adult obese (BMI ≥ 35.0 kg/m2) patients,

Exclusion Criteria:

* type 2 diabetes
* hypertension
* liver or kidney failure
* metabolic syndrome
* taking antinflammatory drugs or dietary supplements
* in the case of women, pregnant or lactating

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Changes in serum triglycerides levels | Within the time of intervention, i. e., 3 months
  A reduction in serum triglycerides of at least 5% of initial concentration

SECONDARY OUTCOMES:
Changes in serum levels of inflammatory proteins, including cytokines | Within the time of intervention, i.e., 3 months
  A reduction in the levels of pro-inflammatory cytokines (IL-6) and adipokines (leptin), and an increase of anti-inflammatory cytokines (IL-10) and adipokines (adiponectin)

OTHER OUTCOMES:
Changes in the Bioenergetic index of PBMNC (monocytes and lymphocytes) | Within the time of intervention, i.e., 3 months
  A change in the amount of energy expended by monocytes and lymphocytes after treatment with omega-3 fatty acids (EPA and DHA)

IPD SHARING:
Plan to Share IPD: Yes
All pertinent data from the participants most likely will be available for their review by Regulatory Authorities, Scientific Committees and other scientific personnel.
Supporting Information: Study Protocol, ICF
Time Frame: After completion of the study
Access Criteria: None assigned